CLINICAL TRIAL: NCT05665595
Title: A Phase 3, Randomized, Double-blind, Active-Comparator-Controlled Clinical Study of Adjuvant MK-7684A (Vibostolimab With Pembrolizumab) Versus Adjuvant Pembrolizumab in Participants With High-risk Stage II-IV Melanoma (KEYVIBE-010)
Brief Title: A Study of Adjuvant Pembrolizumab/Vibostolimab (MK-7684A) Versus Pembrolizumab for Resected High-Risk Melanoma in Participants With High-Risk Stage II-IV Melanoma (MK-7684A-010/KEYVIBE-010)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7684A-010; MK-7684A-010 (Other: MSD); KEYVIBE-010 (Other: MSD); 2022-501417-31-00 (Registry Identifier: EU CT); jRCT2031230099 (Registry Identifier: jRCT); U1111-1280-3661 (Registry Identifier: UTN)
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); T-cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine-based inhibitory motif domains (TIGIT)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab/Vibostolimab (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 17 cycles (up to ~1 year).
  Interventions: Biological: Pembrolizumab/Vibostolimab
- Pembrolizumab (Active Comparator): Participants receive 200 mg pembrolizumab via IV infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 17 cycles (up to ~1 year).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab/Vibostolimab — Co-formulation of pembrolizumab 200 mg/20 mL vial and vibostolimab 200 mg administered as IV infusion for up to 17 administrations
  Other Names: MK-7684A
  Arms: Pembrolizumab/Vibostolimab
Biological: Pembrolizumab — Pembrolizumab 25 mg/mL administered as IV infusion for up to 17 administrations
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab

SUMMARY:
The primary purpose of this study is to compare pembrolizumab/vibostolimab to pembrolizumab with respect to recurrence-free survival (RFS). The primary hypothesis is that pembrolizumab/vibostolimab is superior to pembrolizumab with respect to RFS as assessed by the investigator in participants with high-risk resected Stage IIB, IIC, III and IV melanoma.

DETAILED DESCRIPTION:
With Amendment 4, participants will discontinue treatment with pembrolizumab/vibostolimab.

The protocol-specified futility analysis of the primary outcome measure was completed with a data cut-off of 06-Mar-2024 (Primary Completion Date) and served as the final analysis of the primary outcome measure. Per protocol, 192 participants enrolled after the primary completion date and will be analyzed in the End of Trial analysis.

ELIGIBILITY:
Inclusion Criteria:

* Has surgically resected and histologically or pathologically confirmed diagnosis of Stage IIB and IIC (pathological or clinical), III, or IV cutaneous melanoma per the American Joint Committee on Cancer (AJCC) eighth edition guidelines
* Has not received any prior systemic therapy for melanoma beyond surgical resection
* Has had no more than 12 weeks between final surgical resection and randomization
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on anti-retroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load before randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening

Exclusion Criteria:

* Has ocular, mucosal, or conjunctival melanoma
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has not adequately recovered from major surgical procedure or has ongoing surgical complications
* Has received prior radiotherapy within 2 weeks of start of study intervention or has had a history of radiation pneumonitis
* Received a live or live attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed
* Has received an investigational agent or has used an investigational device within 4 weeks before study intervention administration
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has an active infection requiring systemic therapy
* Has had an allogenic tissue/solid organ transplant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1594 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2025-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (205):
- United States (30):
  - Moores Cancer Center ( Site 0116), La Jolla, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office ( Site 0123), Los Angeles, California
  - UCLA Hematology/Oncology - Westwood (Building 100) ( Site 0131), Los Angeles, California
  - California Pacific Medical Center - Pacific Campus ( Site 0111), San Francisco, California
  - UCSF Medical Center at Mission Bay ( Site 0130), San Francisco, California
  - The Melanoma & Skin Cancer Institute ( Site 0120), Englewood, Colorado
  - Georgetown University Medical Center ( Site 0144), Washington D.C., District of Columbia
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 0110), Miami, Florida
  - Moffitt Cancer Center, Richard M. Shulze Family Foundation Outpatient Center ( Site 0124), Tampa, Florida
  - Northwestern Memorial Hospital ( Site 0109), Chicago, Illinois
  - Advocate Medical Group-Oncology ( Site 0102), Park Ridge, Illinois
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 0107), Iowa City, Iowa
  - Henry Ford Hospital ( Site 0133), Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada ( Site 0142), Las Vegas, Nevada
  - R.J. Zuckerberg Cancer Center-Medical Oncology ( Site 0132), Lake Success, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0146), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center-Hematology and Oncology ( Site 0113), New York, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0118), New York, New York
  - Weill Cornell Medical College ( Site 0115), New York, New York
  - Levine Cancer Institute ( Site 0138), Charlotte, North Carolina
  - Sanford Fargo Medical Center ( Site 0127), Fargo, North Dakota
  - Children's Hospital of Pittsburgh ( Site 0141), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center ( Site 0135), Pittsburgh, Pennsylvania
  - Sanford Cancer Center ( Site 0125), Sioux Falls, South Dakota
  - The West Clinic, PLLC dba West Cancer Center ( Site 0119), Germantown, Tennessee
  - St. Jude Children's Research Hospital ( Site 0106), Memphis, Tennessee
  - Vanderbilt University Medical Center ( Site 0139), Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center ( Site 0145), Houston, Texas
  - Inova Schar Cancer Institute ( Site 0103), Fairfax, Virginia
  - University of Wisconsin Hospital and Clinics ( Site 0108), Madison, Wisconsin
- Argentina (6):
  - Centro de Investigaciones Metabólicas (CINME)-Oncology ( Site 0204), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming-Alexander Fleming ( Site 0209), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC) ( Site 0200), Buenos Aires, Buenos Aires F.D.
  - Instituto de Oncología de Rosario ( Site 0206), Rosario, Santa Fe Province
  - Sanatorio Finochietto ( Site 0212), Buenos Aires
  - Clinica Adventista Belgrano-Oncology ( Site 0211), CABA
- Australia (11):
  - Blacktown Hospital-Blacktown Cancer and Haematology Centre - Medical Oncology ( Site 1464), Blacktown, New South Wales
  - Calvary Mater Newcastle-Medical Oncology ( Site 1462), Waratah, New South Wales
  - Melanoma Institute Australia-Clinical Trials Unit ( Site 1450), Wollstonecraft, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Si, Brisbane, Queensland
  - Cairns Hospital-Clinical Research Unit ( Site 1458), Cairns, Queensland
  - Gallipoli Medical Research Ltd-GMRF CTU ( Site 1451), Greenslopes, Queensland
  - Tasman Oncology Research ( Site 1456), Southport, Queensland
  - Royal Adelaide Hospital-RAH Cancer Centre ( Site 1457), Adelaide, South Australia
  - Icon Cancer Centre Hobart ( Site 1465), Hobart, Tasmania
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 1455), Melbourne, Victoria
  - One Clinical Research ( Site 1460), Nedlands, Western Australia
- Austria (6):
  - Universitätsklinikum St. Pölten-Department of Dermatology ( Site 0606), Sankt Pölten, Lower Austria
  - Medizinische Universität Graz-Innere Medizin Klin. Abt. Onkologie ( Site 0601), Graz, Styria
  - Medizinische Universitaet Innsbruck-Univ Klinik für Dermatologie, Venerologie und Allergologie ( Sit, Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen-Dermatologie ( Site 0602), Linz, Upper Austria
  - Medizinische Universität Wien-Department of Dermatology ( Site 0600), Vienna, Vienna
  - Uniklinikum Salzburg-Department of Dermatology and Allergology ( Site 0604), Salzburg
- Belgium (6):
  - GZA Ziekenhuizen campus Sint-Augustinus ( Site 0655), Wilrijk, Antwerpen
  - Cliniques universitaires Saint-Luc ( Site 0652), Brussels, Bruxelles-Capitale, Region de
  - Jessa Ziekenhuis ( Site 0656), Hasselt, Limburg
  - Université Catholique de Louvain-Namur - Centre Hospitalier -Oncology ( Site 0653), Yvoir, Namur
  - VITAZ-Medical Oncology ( Site 0654), Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven-General Medical Oncology ( Site 0650), Leuven, Vlaams-Brabant
- Brazil (6):
  - Centro Avançado de Tratamento Oncológico- CENANTRON ( Site 0256), Belo Horizonte, Minas Gerais
  - Hospital de Cancer de Londrina-Clinical Research Unit ( Site 0252), Londrina, Paraná
  - Associação Hospitalar Beneficente São Vicente de Paulo-Instituto do Câncer ( Site 0259), Passo Fundo, Rio Grande do Sul
  - ANIMI - Unidade de Tratamento Oncologico ( Site 0255), Lages, Santa Catarina
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia ( Site 0262), Santo André, São Paulo
  - A. C. Camargo Cancer Center ( Site 0258), São Paulo
- Canada (3):
  - The Ottawa Hospital - General Campus-The Ottawa Hospital Cancer Centre ( Site 0004), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 0003), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0006), Toronto, Ontario
- Chile (7):
  - Oncocentro Valdivia ( Site 0307), Valdivia, Los Ríos Region
  - FALP-UIDO ( Site 0303), Santiago, Region M. de Santiago
  - Oncovida ( Site 0304), Santiago, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 0305), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0302), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS-ACEREY ( Site 0300), Viña del Mar, Región de Valparaíso
  - Bradford Hill Norte ( Site 0308), Antofagasta
- China (21):
  - Beijing Ji Shui Tan Hospital ( Site 1657), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Renal carcinoma and melanoma ( Site 1650), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 1651), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 1659), Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center-melanoma ( Site 1655), Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 1668), Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University ( Site 1669), Shijiazhuang, Hebei
  - The Third Hospital of Zhengzhou-Oncology ( Site 1653), Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center-Cancer Center ( Site 1664), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University-Oncology ( Site 1673), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Oncology (, Nanjing, Jiangsu
  - Jiangsu Province Hospital-Oncology Department ( Site 1663), Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 1652), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Oncology ( Site 1665), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 1658), Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital ( Site 1660), Taiyuan, Shanxi
  - West China Hospital, Sichuan University-Head and Neck Oncology ( Site 1667), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital-Biotherapy ( Site 1671), Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi-Bone and Soft Tissue Department ( Site 1674), Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital-Biotherapy Center ( Site 1666), Kunming, Yunnan
  - Zhejiang Cancer Hospital-Oncology ( Site 1661), Hangzhou, Zhejiang
- Colombia (5):
  - Instituto de Cancerología ( Site 0356), Medellín, Antioquia
  - Fundación Colombiana de Cancerología Clínica Vida ( Site 0355), Medellín, Antioquia
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 0358), Bogotá, Bogota D.C.
  - Mediservis del Tolima IPS S.A.S ( Site 0357), Ibagué, Tolima Department
  - Fundación Valle del Lili ( Site 0352), Cali, Valle del Cauca Department
- France (9):
  - Centre Hospitalier de Valence-Service de Dermatologie ( Site 0702), Valence, Drome
  - Hopital Claude Huriez - CHU de Lille-Clinique de Dermatologie ( Site 0700), Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu-Onco-Dermatology ( Site 0707), Nantes, Loire-Atlantique
  - Institut de Cancérologie de l'Ouest-Oncologie Médicale ( Site 0706), Saint-Herblain, Loire-Atlantique
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Ti-Service de Dermatologie et Cancérologi, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de Pau ( Site 0708), Pau, Pyrenees-Atlantiques
  - centre hospitalier lyon sud-Service de dermatologie ( Site 0714), Pierre-Bénite, Rhone
  - Gustave Roussy-Dermatologie ( Site 0713), Villejuif, Val-de-Marne
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 0711), Paris
- Germany (13):
  - Universitaetsklinikum Heidelberg ( Site 0765), Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Mannheim ( Site 0751), Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen-Hautklinik ( Site 0750), Erlangen, Bavaria
  - Klinik und Poliklinik für Dermatologie und Allergologie-Dermato-oncology ( Site 0757), München, Bavaria
  - Elbe Kliniken Stade-Buxtehude, Klinikum Buxtehude-Dermatologisches Zentrum ( Site 0754), Buxtehude, Lower Saxony
  - Medizinische Hochschule Hannover ( Site 0758), Hanover, Lower Saxony
  - Universitaetsklinikum Essen-Klinik für Dermatologie, Venerologie und Allergologie ( Site 0761), Essen, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden-Skin Cancer Center Minden ( Site 0759), Minden, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Dermatologie ( Site 0766), Dresden, Saxony
  - Universitätsklinikum Leipzig ( Site 0762), Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel-Hautklinik ( Site 0767), Kiel, Schleswig-Holstein
  - Charité Universitaetsmedizin Berlin - Campus Mitte-Hauttumorcentrum Charité (HTCC) ( Site 0756), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0752), Hamburg
- India (3):
  - Artemis hospital ( Site 1551), Gurugram, Haryana
  - Tata Memorial Hospital-Medical Oncology ( Site 1550), Mumbai, Maharashtra
  - All India Institute of Medical Sciences-Medical oncology ( Site 1552), New Delhi, National Capital Territory of Delhi
- Ireland (2):
  - St. James's Hospital-Cancer clinical trials office ( Site 0900), Dublin
  - Beaumont Hospital, Dublin-Cancer Clinical Trials & Research Unit ( Site 0902), Dublin
- Israel (6):
  - Emek Medical Center-oncology ( Site 0952), Afula
  - Soroka Medical Center ( Site 0953), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0955), Haifa
  - Hadassah Medical Center ( Site 0951), Jerusalem
  - Rabin Medical Center-Oncology ( Site 0954), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 0950), Ramat Gan
- Italy (9):
  - Instituto Tumori Giovanni Paolo II ( Site 1003), Bari, Apulia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori ( Site 1004), Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1000), Milan, Lombardy
  - A.O.U. Policlinico Paolo Giaccone-Depatment of Discipline Chirurgiche, Oncologiche e Stomatologiche, Palermo, Sicily
  - Azienda Ospedaliero Universitaria Senese ( Site 1005), Siena, Tuscany
  - AO Santa Maria della Misericordia ( Site 1006), Perugia, Umbria
  - Istituto Europeo di Oncologia IRCCS ( Site 1008), Milan
  - Azienda Ospedaliero Universitaria ( Site 1002), Modena
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1001), Napoli
- Japan (6):
  - Nagoya University Hospital ( Site 1753), Nagoya, Aichi-ken
  - Sapporo Medical University Hospital ( Site 1755), Sapporo, Hokkaido
  - Niigata Cancer Center Hospital ( Site 1751), Niigata, Niigata
  - Shizuoka Cancer Center ( Site 1752), Nagaizumi-cho,Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 1750), Chuo-ku, Tokyo
  - Osaka International Cancer Institute ( Site 1754), Osaka
- New Zealand (5):
  - Tauranga Hospital-Bay of Plenty Clinical Trials Unit ( Site 1501), Tauranga, Bay of Plenty
  - New Zealand Clinical Research (Christchurch) ( Site 1509), Christchurch, Canterbury
  - P3 Research - Palmerston North ( Site 1510), Palmerston North, Manawatu-Wanganui
  - Dunedin Hospital ( Site 1511), Dunedin, Otago
  - Harbour Cancer & Wellness ( Site 1508), Auckland
- Poland (11):
  - Szpital Kliniczny im. H. Swiecickiego nr 2-Oddział Kliniczny Onkologii Klinicznej i Doświadczalnej (, Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1061), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow ( Site 1053), Krakow, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1058), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1065), Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Chirurgii Onkologicznej, Transplantacyjnej i Ogólnej ( Site, Gdansk, Pomeranian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. J. Korczaka w Słupsku-Oncologii, Chemioterapii ( Site 1064), Słupsk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 1056), Gliwice, Silesian Voivodeship
  - Zachodniopomorskie Centrum Onkologii ( Site 1063), Szczecin, West Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej ( Site 1054), Kielce, Świętokrzyskie Voivodeship
- South Africa (10):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 1161), Port Elizabeth, Eastern Cape
  - Medical Oncology Centre of Rosebank ( Site 1160), Johannesburg, Gauteng
  - Wilgers Oncology Centre ( Site 1154), Pretoria, Gauteng
  - Curo Oncology ( Site 1158), Pretoria, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 1152), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 1151), Sandton, Gauteng
  - The Oncology Centre ( Site 1157), Durban, KwaZulu-Natal
  - Abraham Oncology ( Site 1150), Richards Bay, KwaZulu-Natal
  - Cape Town Oncology Trials ( Site 1155), Cape Town, Western Cape
  - Cancercare Rondebosch Oncology-Clinical trials ( Site 1159), Rondebosch, Western Cape
- South Korea (3):
  - Seoul National University Hospital-Oncology ( Site 1600), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1601), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 1602), Seoul
- Spain (6):
  - Institut Català d'Oncologia - L'Hospitalet ( Site 1202), L'Hospitalet de Llobregat, Barcelona
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 1203), Doniostia - San Sebastian, Gipuzkoa
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 1204), Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital General-Oncology ( Site 1201), Málaga, Malaga
  - Hospital General Universitario de Valencia ( Site 1200), Valencia, Valenciana, Comunitat
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 1205), Seville
- Sweden (2):
  - Länssjukhuset Ryhov-Onkologkliniken ( Site 1253), Jönköping, Jönköping County
  - Karolinska Universitetssjukhuset Solna ( Site 1252), Stockholm, Stockholm County
- Switzerland (8):
  - University Hospital Basel ( Site 1303), Basel, Canton of Basel-City
  - Inselspital Bern ( Site 1301), Bern, Canton of Bern
  - Hôpitaux Universitaires de Genève (HUG)-Oncology ( Site 1307), Geneva, Canton of Geneva
  - CHUV (centre hospitalier universitaire vaudois) ( Site 1304), Lausanne, Canton of Vaud
  - UniversitätsSpital Zürich-Dermatology ( Site 1300), Zürich Flughafen, Canton of Zurich
  - Ospedale Regionale Bellinzona e Valli ( Site 1308), Bellinzona, Canton Ticino
  - Hôpital de Sion ( Site 1305), Sion, Valais
  - Cantonal Hospital St.Gallen-Oncology & Hematology ( Site 1306), Sankt Gallen
- Turkey (Türkiye) (8):
  - Ankara City Hospital-Medical Oncology ( Site 1357), Çankaya, Ankara
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 1360), Izmir, Karsiyaka, İzmir
  - Hacettepe Universite Hastaneleri ( Site 1363), Ankara
  - Liv Hospital Ankara-Oncology ( Site 1353), Ankara
  - Akdeniz Universitesi Hastanesi-Medical Oncology ( Site 1355), Antalya
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1358), Istanbul
  - Mersin Sehir Eğitim ve Araştırma Hastanesi-Oncology ( Site 1361), Mersin
  - Ondokuz Mayıs Universitesi-Oncology department ( Site 1359), Samsun
- United Kingdom (3):
  - Addenbrooke's Hospital ( Site 1400), Cambridge, Cambridgeshire
  - University College London Hospital ( Site 1405), London, England
  - Guy's & St Thomas' NHS Foundation Trust-Oncology & Haematology Clinical Trials ( Site 1401), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Shapira-Frommer R, Niu J, Perets R, Peters S, Shouse G, Lugowska I, Garassino MC, Sands J, Keenan T, Zhao B, Healy J, Ahn MJ. The KEYVIBE program: vibostolimab and pembrolizumab for the treatment of advanced malignancies. Future Oncol. 2024;20(27):1983-1991. doi: 10.1080/14796694.2024.2343272. Epub 2024 Sep 4. PMID 39230120
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26262&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol-specified final analysis for the following results, including the participant flow, was performed on 1402 participants that enrolled within the primary completion data cut-off. Analysis of the remaining 192 enrolled participants will be included in the End of Trial analysis.
Groups:
- Pembrolizumab/Vibostolimab: Participants received pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 17 cycles (up to ~1 year).
- Pembrolizumab: Participants received 200 mg pembrolizumab via IV infusion on Day 1 of each cycle (cycle length = 3 weeks) for up to 17 cycles (up to ~1 year).
Period: Overall Study
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab
Started | 701 | 701
Treated | 698 | 700
Completed | 0 | 0
Not Completed | 701 | 701
Not completed — Ongoing | 692 | 698
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 6 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol, analysis population consisted of all participants randomized by the primary completion data cut-off.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab | Total
Number analyzed (Participants) | 701 | 701 | 1402
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (13.8) | 59.2 (13.9) | 59.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 291 | 573
  Male | 419 | 410 | 829
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 73 | 157
  Not Hispanic or Latino | 585 | 586 | 1171
  Unknown or Not Reported | 32 | 42 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 134 | 139 | 273
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 3 | 2 | 5
  White | 553 | 554 | 1107
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 2 | 1 | 3
Risk-based Melanoma Stage [Count of Participants; unit: Participants] — Participants were stratified by melanoma stage using the American Joint Committee on Cancer (AJCC) 8th edition: Stage IIB/IIC/clinical IIB and IIC/IIIA/IIIB versus Stage IIIC/IIID/IV. Stage IIB (primary tumor [PT] >2mm), Stage IIC (>4mm PT + ulceration), Stage IIIA (<1mm PT and 1-3 positive sentinel lymph node [LN+]), Stage IIIB (No evidence of PT; <4mm PT AND 1-3 LN+ or microsatellite metastases [SM]), Stage IIIC (0mm PT AND 2-3 LN+; <2-4mm PT +/- ulceration and SM and/or >1 LN+; 0-2mm PT and >2 LN+), Stage IIID (>4mm PT ulceration and >2 LN+ and SM), Stage IV (Evidence of distant metastases)
  Participants
    Stage IIB/IIC/clinical IIB and IIC/IIIA/IIIB | 427 | 427 | 854
    Stage IIIC/IIID/IV | 274 | 274 | 548
Region of Enrollment [Count of Participants; unit: Participants] — Participants were stratified by region of enrollment; Asia versus Rest of the World (ROW).
  Participants
    Asia | 133 | 135 | 268
    Rest of the World (ROW) | 568 | 566 | 1134

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-Free Survival (RFS)
Description: RFS is defined as the time from randomization to any recurrence (local, locoregional, regional, or distant) as assessed by the investigator, or death due to any cause, whichever occurs first. The RFS as assessed by the investigator is presented for all randomized participants. Protocol pre-specified final analysis for this outcome measure was conducted with the primary completion data cut-off.
Time Frame: Up to approximately 13 months
Population: Per protocol, analysis population consisted of all participants randomized, by the primary completion data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab
Number analyzed (Participants) | 701 | 701
Months | NA [NA to NA] — Median, upper limit, and lower limit not reached at the time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median, upper limit, and lower limit not reached at the time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab/Vibostolimab vs Pembrolizumab; Test type: Other; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.87 to 1.80] — Hazard Ratio based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by melanoma risk-based stage (IIB/IIC/clinical IIB and IIC/IIIA/IIIB vs IIIC/IIID/IV) and region of enrollment (Asia vs ROW)

2. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 31 months
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 31 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 13 months
Description: All-cause mortality: all participants randomized by the primary completion data cut-off. AEs: all participants randomized by the primary completion data cut-off who received ≥1 dose of treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression (NP)", "Malignant NP" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 6/701 | 1/701
Serious Adverse Events (participants affected / at risk) | 109/698 | 57/700
Other Adverse Events (participants affected / at risk) | 462/698 | 426/700
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab (N=698) | Pembrolizumab (N=700)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 6 (6) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal disorder (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 14 (14) | 2 (2)
Hypophysitis (Endocrine disorders) | 5 (5) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Immune-mediated hypophysitis (Endocrine disorders) | 2 (2) | 0 (0)
Immune-mediated hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Optic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vogt-Koyanagi-Harada disease (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 4 (4) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 5 (5) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 1 (1)
Meningitis aseptic (Infections and infestations) | 3 (3) | 0 (0)
Meningoencephalitis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin graft necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Persistent postural-perceptual dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab (N=698) | Pembrolizumab (N=700)
Hyperthyroidism (Endocrine disorders) | 88 (97) | 80 (82)
Hypothyroidism (Endocrine disorders) | 66 (67) | 64 (65)
Diarrhoea (Gastrointestinal disorders) | 66 (80) | 71 (89)
Nausea (Gastrointestinal disorders) | 47 (55) | 58 (73)
Asthenia (General disorders) | 35 (42) | 19 (21)
Fatigue (General disorders) | 131 (148) | 144 (166)
Alanine aminotransferase increased (Investigations) | 68 (79) | 69 (80)
Aspartate aminotransferase increased (Investigations) | 64 (73) | 52 (60)
Arthralgia (Musculoskeletal and connective tissue disorders) | 75 (97) | 69 (80)
Headache (Nervous system disorders) | 61 (70) | 48 (58)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (45) | 34 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 178 (202) | 91 (100)
Rash (Skin and subcutaneous tissue disorders) | 167 (194) | 76 (91)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 48 (57) | 22 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT05665595/Prot_SAP_000.pdf